CLINICAL TRIAL: NCT01612923
Title: Safety and Efficacy of Medical Abortion Provided by Midlevel Providers or Physicians
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kristina Gemzell Danielsson (Other)
Responsible Party: Sponsor-Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W2010U
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2012-06

CONDITIONS: Medical Abortion
Keywords: abortion; medical abortion
MeSH Terms: interventions — Nurse Midwives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midwife (Experimental): Gynecological exam and ultrasound performed by midwife, medical abortion service provided by midwife,contraceptive advice provided by midwife. Follow-up visit provided by midwife
  Interventions: Other: Midwife
- Physician (No Intervention): Gynecological exam and ultrasound and contraceptive advice provided by physician. Medical abortion service and follow-up visit provided by midwife

INTERVENTIONS:
Other: Midwife — gynecological exam and ultrasound and contraceptive advice provided by midwife
  Arms: midwife

SUMMARY:
The physical examination before an abortion is usually performed by a physician. However, in many countries access to physicians is limited. To increase access to safe abortion this study wishes to examine if midlevel providers such as specially trained midwives can provide safe abortion services. Midwives in study were specially trained to perform early pregnancy ultrasound and if needed to consult a physician. The midwife then provided the abortion service as well as the contraceptive advice. Women were randomized to receive the service from a midwife or a physician.

ELIGIBILITY:
Inclusion Criteria:

* healthy women aged 18-45 with no contraindication to medical abortion

Exclusion Criteria:

* any medical condition which contraindicates medical abortion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1180 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
feasibility | 3 weeks
  Successful completion of abortion without need for unscheduled visits or calls.

SECONDARY OUTCOMES:
efficacy | 3 weeks
  complete uterine evacuation without the need for further medical or surgical intervention
acceptability | 3 weeks
  as assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell Danielsson, professor, Principal Investigator — Karolinska Institutet; Helena Kopp Kallner, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Kopp Kallner H, Gomperts R, Salomonsson E, Johansson M, Marions L, Gemzell-Danielsson K. The efficacy, safety and acceptability of medical termination of pregnancy provided by standard care by doctors or by nurse-midwives: a randomised controlled equivalence trial. BJOG. 2015 Mar;122(4):510-7. doi: 10.1111/1471-0528.12982. Epub 2014 Jul 18. PMID 25040643